CLINICAL TRIAL: NCT00440063
Title: A Randomized Study to Compare the Safety and Effectiveness of Two Monitoring Schedules to Maintain Hemoglobin Levels and Iron Parameters in Patients With Renal Anemia Receiving NeoRecormon
Brief Title: A Study of NeoRecormon (Epoetin Beta) in Patients With Renal Anemia.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20828
Record Dates: First submitted 2007-02-23; First posted 2007-02-26 (Estimated); Last update posted 2007-12-20 (Estimated); Status verified 2007-12

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — epoetin beta

INTERVENTIONS:
Drug: epoetin beta [NeoRecormon]

SUMMARY:
This study will determine whether 8 weekly monitoring of hemoglobin and iron parameters in the correction phase of NeoRecormon therapy in patients with renal anemia is as safe and effective as 4 weekly monitoring. Patients with chronic kidney disease will receive NeoRecormon at a dose aimed at achieving and maintaining a Hb level of 110-130g/L. They will be randomized into one of two schedules for monitoring hemoglobin levels and iron parameters, either 4 weekly or 8 weekly. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 inidividuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-80 years of age;
* stage 3-4 chronic kidney disease (eGFR 15-60mL/min);
* Hb <100g/L, TSAT>=20%, and ferritin >=100 mcg/L at screening.

Exclusion Criteria:

* anticipating to go on renal replacement therapy;
* anticipating a living related-donor kidney transplant, or a prior recipient of a kidney transplant;
* uncontrolled hypertension;
* congestive heart failure;
* active bleeding or red blood cell transfusions in 8 weeks prior to screening; systematic hematological disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Percentage of patients achieving target Hb within 20 weeks.

SECONDARY OUTCOMES:
Efficacy: % of patients exceeding upper Hb target; % who fail to reach target Hb; median time to achieve Hb target; dose of NeoRecormon required to meet target Hb concentration; % who maintain target iron parameters. Safety: AEs, SAEs.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- Australia (9):
  - Adelaide
  - Gosford
  - Herston
  - Liverpool
  - Parkville
  - Perth
  - Sydney
  - Tasmania
  - Woolloongabba